CLINICAL TRIAL: NCT02910375
Title: A Prospective Multi-centric Belgian Trial to Validate the Use of Golimumab Serum Level Analysis Using the Dried Blood Spot (DBS) Methodology
Brief Title: Golimumab Dried Blood Spot Analysis
Acronym: GOUDA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: General Hospital Groeninge (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S59372
Record Dates: First submitted 2016-09-12; First posted 2016-09-22 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Ulcerative Colitis
Keywords: golimumab; drug monitoring; home based care
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Other): Patients starting golimumab therapy Week 0: 200 mg Week 2: 100 mg Week 6, 10, 14, and 18: 50 mg (<80 kg) or 100mg (>80 kg body weight)
  Interventions: Other: Cohort A
- Cohort B (Other): Patients already on golimumab therapy will continue their actual treatment 50 mg every 4 weeks (<80 kg) or 100mg every 4 weeks (>80 kg body weight)
  Interventions: Other: Cohort B

INTERVENTIONS:
Other: Cohort A — Venous sampling (n=13) will be performed in the hospital at D0 (prior to first golimumab injection), D3, D7, D14 (prior to second injection), D28, M0D0 (right before injection at week 6), M0D3, M0D7, M1D0 (4 weeks after M0D0, week 10), M1D3, M1D7, M2D0 (8 weeks after M0D0, week 14), M3D0 (12 weeks after M0D0, week 18) Dried blood spot sampling (n=39) will be performed at D0 (prior to first golimumab injection), D1, D2, D3, D4, D5, D6, D7, D10, D14, D15, D16, D17, D18, D19, D20, D21, D28, D35, M0D0 (right before injection at week 6), M0D3, M0D7, M1D0 (4 weeks after M0D0, week 10), M1D1, M1D3, M1D5, M1D7, M1D9, M1D14, M1D21, M2D0 (8 weeks after M0D0, rig week 14), M2D1, M2D3, M2D5, M2D7, M2D9, M2D14, M2D21, M3D0 (12 weeks after M0D0, week 18)
  Other Names: Monitoring through serum and dry blood spot analysis
  Arms: Cohort A
Other: Cohort B — Venous sampling (n=8) will be performed at M0D0 (right before new golimumab injection), M0D3, M0D7, M1D0 (4 weeks after M0D0, right before next injection), M1D3, M1D7, M2D0 (8 weeks after M0D0, right before next injection), M3D0 (12 weeks after M0D0, right before next injection) Dried blood spot sampling (n=20) will be performed at M0D0 (right before new golimumab injection), M0D3, M0D7, M1D0 (4 weeks after M0D0, right before next injection), M1D1, M1D3, M1D5, M1D7, M1D9, M1D14, M1D21, M2D0 (8 weeks after M0D0, right before next injection), M2D1, M2D3, M2D5, M2D7, M2D9, M2D14, M2D21, M3D0 (12 weeks after M0D0, right before next injection)
  Other Names: Monitoring through serum and dry blood spot analysis
  Arms: Cohort B

SUMMARY:
This retrospective multi-centric Belgian prospective trial will involve 10 patients initiating or under maintenance subcutaneous golimumab therapy for moderate-to-severe colitis at the University Hospitals Leuven (Leuven, Belgium) or AZ Groeninge (Kortrijk, Belgium)

Patients will (have) receive(d) standard induction therapy with golimumab 200mg at week 0, and golimumab 100mg at week 2. Maintenance therapy will (have) start(ed) at week 6, with 50 or 100mg of golimumab every 4 weeks, depending on body weight (50mg every 4 weeks for patients with a body weight of less than 80kg, and 100mg for the others)

Patients will come to the hospital for clinical evaluation, blood sampling and golimumab administration following daily clinical practice. The patients will be requested to perform several dry blood spot analyses at home.

DETAILED DESCRIPTION:
BLOOD SAMPLING:

Blood samples are collected using two sampling methods at different time points (indicated on the timeline above); DBS sampling (max 39 samples/patient) and venous blood sampling (max 13 samples/patient). Venous blood sampling will be performed during a standard outpatient clinic in one of the participating centres, and forwarded to the Laboratory for Therapeutic and Diagnostic Antibodies in Leuven for further analyses. DBS samples will be send directly to the Laboratory for Therapeutic and Diagnostic Antibodies in Leuven through classical mailing.

DBS sampling will be performed by the patient during the outpatient clinic (at same moment as venous punctures, max 13 samples/patient) and at home for the intermediate values (max 26 samples/patient). Patients will be taught how to perform a finger prick during the outpatient clinic. A conversion factor will be defined. Determination of concentration-time profile and exposure of golimumab in the individual patients will be performed by intensive sampling for 3 to 4.5 months. Time point of max concentration, intermediate concentration, and trough concentration will be determined in each patient.

Note: A similar procedure will be adopted to measure free anti-golimumab antibody concentrations on the DBS using a drug sensitive assay. Free anti-golimumab antibody concentrations will be measured when the serum golimumab concentration is below limit of quantification.

MEASUREMENT OF GOLIMUMAB AND ANTI-GOLIMUMAB ANTIBODY CONCENTRATIONS:

Golimumab concentrations will be measured using a sandwich type ELISA, in which golimumab is captured between an immobilized monoclonal antibody towards golimumab (MA-GLM) 171D8 and an added horseradish peroxidase (HRP)-labeled MA-GLM159B8. The assay was developed and validated, analytically (external and internal) and clinically, as described by Detrez et al. Golimumab concentrations will be measured on every sample.

Free anti-golimumab antibody concentrations will be measured using a drug sensitive assay. Total anti-golimumab antibody concentrations will be measured using a drug tolerant assay. Development and validation (analytical + clinical) of these assays is described by Detrez et al. Total anti-golimumab antibody concentrations will be measured on every venous sample. Free anti-golimumab antibody concentrations will be measured when the serum golimumab concentration is below limit of quantification on both venous sample and DBS sample (based on adalimumab serum concentrations measured in by our laboratory, we expect that 11% of samples measured within the first year of treatment have an undetectable golimumab concentration).

BASELINE CHARACTERISTICS:

* Baseline characteristics will include: sex, age at diagnosis, weight, body mass index, disease extent, smoking status (never, ex, active), primary sclerosing cholangitis, haemoglobin, serum albumin, and C-reactive protein
* Previous medical characteristics will include previous use of mesalamine, steroids, immunosuppressive agents, ciclosporin, infliximab, adalimumab, vedolizumab, …
* Current medical characteristics will include use of mesalamine, use of steroids (dosing, duration since initiation), use of immunosuppressive agents (dosing, duration since initiation), use of golimumab (dosing, duration since initiation, last dose), …

QUESTIONNAIRE REGARDING PATIENT FRIENDLINESS:

• At the end of the study the participants will be requested to fill out a questionnaire regarding the patient friendliness of the dried blood spot (DBS) methodology

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 at moment of inclusion
* Established diagnosis of ulcerative colitis (UC)
* Patients under golimumab therapy for moderate-to-severe colitis, including minimally 3 patients who will initiate golimumab therapy

Exclusion Criteria:

* Subjects with Crohn's disease, or IBD type unclassified
* Subjects who underwent a subtotal colectomy or proctocolectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of golimumab serum sample through venous puncture and dried blood spot analysis | During 4.5 months for golimumab starters and 3.0 months for patients under golimumab maintenance therapy
  The primary objective of this prospective multi-centric Belgian trial is to compare golimumab serum concentrations obtained using venous puncture, with golimumab serum concentrations obtained using DBS sampling and extraction, and to determine its robustness

SECONDARY OUTCOMES:
Area under the curve of golimumab exposure during induction therapy | 1.5 months
  To determine the area under the curve of golimumab exposure in individual patients with moderate to severe colitis initiating golimumab therapy, by frequent analysis of golimumab serum levels using dried blood spot analysis
Area under the curve of golimumab exposure during maintenance therapy | 3.0 months
  To determine the area under the curve of golimumab exposure in individual patients with moderate to severe colitis under maintenance therapy with golimumab by frequent analysis of golimumab serum levels using dried blood spot analysis
Maximum golimumab serum concentration during induction therapy | 1.5 months
  To determine the timing of the maximum golimumab concentration in individual patients with moderate to severe colitis initiating golimumab therapy by frequent analysis of golimumab serum levels using dried blood spot analysis
Maximum golimumab serum concentration during maintenance therapy | 3.0 months
  To determine the timing of the maximum golimumab concentration in individual patients with moderate to severe colitis under maintenance therapy with golimumab by frequent analysis of golimumab serum levels using dried blood spot analysis
Patient perception question 1: The information I received from my physician and colleagues regarding dried blood spot analyses was adequate | After 4.5 months for golimumab starters and after 3.0 months for patients under golimumab maintenance therapy
  Score to check for adequate information. Possible answers: certainly not, no, I don't know, yes, for sure
Patient perception question 2: I had fluent access to further information on all aspects of the dried blood spot analysis | After 4.5 months for golimumab starters and after 3.0 months for patients under golimumab maintenance therapy
  Score to check for accessibility for extra help. Possible answers: certainly not, no, I don't know, yes, for sure
Patient perception question 3: With the provided tools it was easy to get a blood spot on the paper. | After 4.5 months for golimumab starters and after 3.0 months for patients under golimumab maintenance therapy
  Score to check for easiness of getting blood spot. Possible answers: certainly not, no, I don't know, yes, for sure
Patient perception question 4: With the provided tools it was easy to send/bring the paper with the dried blood spot to the physician/lab | After 4.5 months for golimumab starters and after 3.0 months for patients under golimumab maintenance therapy
  Score to check for easiness of getting paper with dried blood spot to the physician/lab. Possible answers: certainly not, no, I don't know, yes, for sure
Patient perception question 5: I prefer to perform the dried blood spot at home than to go to the hospital for venous sampling | After 4.5 months for golimumab starters and after 3.0 months for patients under golimumab maintenance therapy
  Score to check for preference of dried blood spot analysis over venous sampling. Possible answers: certainly not, no, I don't know, yes, for sure
Patient perception question 6: In general this dried blood spot system is user friendly | After 4.5 months for golimumab starters and after 3.0 months for patients under golimumab maintenance therapy
  Score to check for userfriendliness of dried blood spot analysis. Possible answers: certainly not, no, I don't know, yes, for sure

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ferrante, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (2):
- Belgium (2):
  - AZ Groeninge, Belgium, Kortrijk
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Detrez I, Schops G, Lefrere J, Tops S, Van Assche G, Vermeire S, Van Moerkercke W, Ferrante M, Gils A. Golimumab Dried Blood Spot Analysis (GOUDA): a Prospective Trial Showing Excellent Correlation with Venepuncture Samples and More Detailed Pharmacokinetic Information. AAPS J. 2018 Dec 18;21(1):10. doi: 10.1208/s12248-018-0282-x. PMID 30564993